CLINICAL TRIAL: NCT06152770
Title: Comparison of Turkish Children's Actual Weights With Predicted Weights Values by APLS, Luscombe and Owens, Best Guess, Nelson Formulas and Broselow Band Methods
Brief Title: Comparison of Turkish Children's Actual Weights With Which Predicted Weights by Estimation Methods
Acronym: CTCAWPWM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Yesim Senayli, assistant professor, Bozok University
Other Study IDs: YSenayli
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Pediatric Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to compare body weigth with the prediceted weigth values abtracted by weigth estimation methods in Turkish Children.

The main question it aims to answer is: to evaluate the suitability of APLS, Luscombe & Owens, Best Guess, Nelson Formula and Broselow Band methods in estimating actual measurements in patients coming to the surgery outpatient clinic of our hospital

ELIGIBILITY:
Inclusion Criteria:admitted to the pediatric surgery clinic 0-18 years old patients will be included

Exclusion Criteria:Those who have a disease that will cause severe developmental growth retardation will be excluded

Ages: 0 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients between the ages of 0-18 who applied to the pediatric surgery outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of actual weigth with predicted weigth | one year

IPD SHARING:
Plan to Share IPD: Undecided